CLINICAL TRIAL: NCT06336954
Title: Exploratory Study of Adibelimab Combined With Famitinib and Chemotherapy for the Treatment of Patients With Driver Gene-Negative Locally Advanced or Metastatic NSCLC Progressing After PD-1 Monoclonal Antibody Combined With Chemotherapy
Brief Title: Adibelimab, Famitinib and Chemotherapy for Advanced NSCLC After PD-1 Inhibitor Failure
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-NSCLC-#-037
Record Dates: First submitted 2024-03-19; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — famitinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Adibelimab (1200mg, IV, every 3 weeks) combined with Famitinib (20mg, daily, orally) and Albumin-bound Paclitaxel (260mg/m2, Day 1, every 3 weeks).
  Interventions: Drug: Adibelimab

INTERVENTIONS:
Drug: Adibelimab — Adibelimab (1200mg, IV, every 3 weeks) combined with Famitinib (20mg, daily, orally) and Albumin-bound Paclitaxel (260mg/m2, Day 1, every 3 weeks)
  Other Names: Famitinib; Chemotherapy

SUMMARY:
This prospective, single-arm trial explores the efficacy of Adibelimab monoclonal antibody combined with Famitinib and chemotherapy in treating locally advanced or metastatic NSCLC patients with negative driver genes who have progressed after PD-1 monoclonal antibody and chemotherapy treatment. The study focuses on assessing progression-free survival (PFS) in 40 participants. Key objectives include evaluating PFS and understanding the progression patterns post-first-line immunotherapy, with an interest in whether switching from PD-1 to PD-L1 inhibitors can overcome immune resistance.

DETAILED DESCRIPTION:
This study is a prospective, single-arm clinical investigation. It aims to assess the effectiveness of the Adibelimab monoclonal antibody in combination with Famitinib and chemotherapy for treating patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) without driver mutations, who have progressed following initial treatment with PD-1 monoclonal antibodies and chemotherapy. The study's primary focus is on evaluating progression-free survival (PFS) among the 40 participants, spanning from December 2023 to December 2026. It intends to explore the therapeutic potential of switching from PD-1 to PD-L1 inhibitors in overcoming immune resistance and identify subgroups that may particularly benefit from this treatment strategy, thereby providing insights into personalized therapy for advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be adults (≥18 years) who have signed an informed consent form.
* They should have an ECOG performance status of 0-1. Diagnosed with stage IIIB-IV NSCLC and have progressed after PD-1 inhibitor treatment.
* Expected to live at least 3 months and have at least one measurable lesion per RECIST v1.1.
* Laboratory test results must meet specific criteria for blood counts, liver and kidney function, and coagulation parameters.
* Patients with stable, treated brain metastases are eligible.
* Women of childbearing potential and men with partners of childbearing potential must agree to use contraception.

Exclusion Criteria:

* Prior therapy with anti-PD-L1, anti-PD-L2, other immune checkpoint inhibitors, or specific cancer treatments.
* Certain cancer types, known mutations, or recent use of systemic corticosteroids or immunosuppressive medications.
* Active brain or leptomeningeal metastases without stability post-treatment, recent severe infections, or major surgery.
* Other conditions that might interfere with the study, such as uncontrollable third-space fluid accumulations, active autoimmune diseases or infections, significant bleeding or thromboembolic events, serious heart conditions, severe allergies to study drugs, other active malignancies, HIV/AIDS, hepatitis B or C infection, or participation in another interventional clinical study within a specified period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival time (PFS) | 4 months
  the time from the start of the first dose of medication to the first occurrence of disease progression (as confirmed by the researcher according to RECIST v1.1 standards) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate | 4 months
  Objective Response Rate
Duration of Response | 4 months
  Duration of Response
Overall Survival | 4 months
  Overall Survival
Treatment-Related Adverse Events | 4 months
  Incidence rates of Treatment-Related Adverse Events, Serious Adverse Events and Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Hui Guo, Principal Investigator — Second Affiliated Hospital of Xian Jiaotong University